CLINICAL TRIAL: NCT04294056
Title: A Single-center, Open-label, Randomized, Two-stage, Two-way Crossover Study to Evaluate the Differences in Pharmadynamics, Pharmacokinetics, and Safety Between Ciprofol and Propofol at Different Doses in Healthy Subjects
Brief Title: A Study to Evaluate the Differences in Pharmadynamics, Pharmacokinetics, and Safety Between Ciprofol and Propofol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-109
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol (Experimental): First-stage: 0.4mg/kg, 0.6 mg/kg, 0.8 mg/kg Second-stage: 0.4mg/kg, 0.6 mg/kg, 0.8 mg/kg
  Interventions: Drug: Ciprofol
- Propofol (Active Comparator): First-stage: 2.0mg/kg, 3.0 mg/kg, 4.0 mg/kg Second-stage: 2.0mg/kg, 3.0 mg/kg, 4.0 mg/kg
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — First-stage: 0.4mg/kg, 0.6 mg/kg, 0.8 mg/kg Second-stage: 0.4mg/kg, 0.6 mg/kg, 0.8 mg/kg
  Arms: Ciprofol
Drug: Propofol — First-stage: 2.0mg/kg, 3.0 mg/kg, 4.0 mg/kg Second-stage: 2.0mg/kg, 3.0 mg/kg, 4.0 mg/kg
  Arms: Propofol

SUMMARY:
This is a single-center, open-label, randomized, two-stage, two-way crossover Phase I study in healthy male subjects.The main objective is to evaluate the differences in pharmadynamics (PD), pharmacokinetics (PK), and safety between ciprofol injectable emulsion and propofol injectable emulsion at different doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males, aged 18-45 years (inclusive);
2. Body weight ≥ 50 kg, body mass index (BMI) between 18-26 kg/m^2 (inclusive);
3. Blood pressure between 90-140/50-90 mmHg (inclusive); heart rate between 60-100 bpm (inclusive); body temperature between 35.4-37.5°C (inclusive); respiratory rate between 12-20 breaths per min (inclusive); SpO2 when inhaling ≥ 92%;
4. Normal results of physical examination, laboratory tests (routine blood, routine urine, blood biochemistry (including hepatic function, renal function, blood glucose, and electrolytes such as Na, K, and Mg), and blood coagulation), 12-lead ECG, and abdominal ultrasonography, or abnormalities considered by the investigators to be clinically insignificant; no significant potential difficult airway (modified Mallampati score Class I-II);
5. No previous history of primary diseases in major organs, such as liver, kidneys, digestive tract, blood, and metabolic diseases; no history of malignant hyperthermia and other hereditary disorders; no history of mental/neurological disorders; no history of epilepsy; no contraindications for deep sedation/general anesthesia; no clinically significant history of anesthesia accidents;
6. Subjects must understand the procedures and methods of this study, and be willing to signing the informed consent form and to complete the trial in strict accordance with clinical trial protocol;

Exclusion Criteria:

1. Patients with known allergies to ciprofol injectable emulsion, excipient in propofol injectable emulsion (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate, and sodium hydroxide); history of drug allergies (including other anesthetics), allergic diseases, or hyperactive immune response;
2. Patients receiving any of the following drugs or therapies prior to screening/administration:

   1. History of drug abuse within 3 months prior to screening, or positive result in urine drug screening during baseline period;
   2. Participated in other drug/medical device trials within 3 month prior to screening;
   3. Serious infection, trauma, or major surgery within 4 weeks prior to screening.
   4. Acute disease with clinical significance (determined by the investigators) within 2 weeks prior to screening, including GI diseases or infections (such as respiratory tract or CNS infections);
   5. Patients who received propofol, other sedatives/anesthetics, and/or opioid analgesics within 1 week prior to administration;
   6. Patients who received prescription drugs, Chinese herbal medicines, over-the-counter drugs, or food supplements (such as vitamins and calcium supplements) other than contraceptives, paracetamol, oral non-steroidal anti-inflammatory drugs, and topical over-the-counter preparations, within 2 weeks prior to administration; those who received UGT or CYP2B6 inhibitors within 7 days prior to administration (refer to Attachment 6 for prohibited drugs); patients can only be enrolled when the principal investigator (PI) and the sponsor agree that the medication has no effect on the safety and PK/PD results of the trial;
3. Patients with history or evidence of any of the following diseases prior to screening/administration:

   1. History of cardiovascular diseases, such as postural hypotension, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction within 6 months before screening, tachycardia/bradycardia requiring medications, third-degree atrioventricular block, or QTcF interval ≥ 450 ms (per Fridericia's correction formula);
   2. Subjects with hypopnea, history of obstructive pulmonary disease, history of asthma, or sleep apnea syndrome; subjects with history of failed endotracheal intubation; history of bronchospasm requiring interventions within 3 months prior to screening; acute upper respiratory tract infection within 1 week prior to baseline, with symptoms such as fever, wheeze, nasal obstruction, or cough;
   3. History of gastrointestinal disorders: history of gastrointestinal retention, active hemorrhage, or conditions that may lead to reflux and aspiration;
4. Laboratory results meeting any of the following during screening/at baseline:

   1. Positive result for any of the markers, including HBsAg, HCV-Ab, HIV-Ab, and Tp-Ab;
   2. Results for hepatic and renal functions exceeding the following ranges:

   ALT or AST > 50% of ULN; Creatinine > 20% of ULN; Total bilirubin > 40% of ULN.
5. History of alcohol abuse within 3 months prior to screening; alcohol abuse defined as average of > 2 units of alcohol per day (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine), or positive alcohol breath test results at baseline;
6. Patients who smoked more than 5 cigarettes per day and a total of more than 60 cigarettes within 3 months prior to screening;
7. Blood donation or blood loss ≥ 200 mL within 30 days prior to screening; plasma donation or plasma exchange within 7 days prior to screening;
8. Subjects who consumed any beverages or foods containing alcohol, grapefruit juice or methylxanthine (such as coffee, tea, cola, chocolate, and energy drinks), participated in strenuous physical activities and had other factors that may affect drug absorption, distribution, metabolism, and excretion, within 2 days prior to baseline; subjects who were unable to fast for 8 hours before dose administration;
9. Subjects who were expected to go through surgery or hospitalization during the trial;
10. Subjects unsuitable for arterial blood collection, such as subjects with positive results in Allen's test;
11. Subjects who were unwilling to practice contraception during the trial; subjects who were planning to conceive within 3 month after the completion of the trial;
12. Subjects judged by the investigators to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Modified observer's assessment of alertness/sedation（MOAA/S） | From first dose of study drug until fully alert on day 1
  Observe the change of modified observer's assessment of alert /sedation during the whole trial
Bispectral index （BIS） | From first dose of study drug until fully alert on day 1
Safety by measurement of Adverse Events | First dose of study drug on day 1

SECONDARY OUTCOMES:
Peak concentration (Cmax) | First dose of study drug on day 1
Area under the plasma concentration versus time curve (AUC) | First dose of study drug on day 1
Terminal half-life (t1/2) | First dose of study drug on day 1
time to peak concentration (Tmax) | First dose of study drug on day 1
clearance (CL) | First dose of study drug on day 1
mean residence time (MRT) | First dose of study drug on day 1
volume of distribution (Vz) | First dose of study drug on day 1

OTHER OUTCOMES:
Use of dynamometer to estimate Muscular strength of lower limbs | From 30 minutes before administration to 1 hour after administration on day 1
The differences between the Montreal Cognitive Assessment (MoCA) test score in Ciprofol group and in a control group of Propofol | From the baseline period to 1 hour after administration on day 1
  Total score of the MoCA,the higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, China